CLINICAL TRIAL: NCT04483102
Title: A Prospective, Single-Center, Non-Randomized, Clinical Trial of Transplantation of Discarded Livers Using Normothermic Machine Perfusion (NMP)
Brief Title: RESTORE Declined Livers Study
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: Mid-America Transplant (Other); OrganOx Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 202007093
Record Dates: First submitted 2020-07-14; First posted 2020-07-23 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-06

CONDITIONS: Liver Diseases; Surgery; Transplant; Failure, Liver
MeSH Terms: conditions — Liver Diseases

STUDY DESIGN:
Intervention Model Description: To successfully transplant NMP-treated livers to patients that would otherwise have been discarded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Declined liver in Normothermic Machine Perfusion (NMP) (Experimental): The discarded livers rejected by all other centers and meeting pre-NMP eligibility criteria will receive NMP using the OrganOx® metra device. The NMP-treated liver that meets the viability criteria will be transplanted to patients who are eligible and consented to the study. NMP of the donated declined liver utilizing the OrganOx® metra device. NMP involves (warm) machine perfusion with oxygenated blood at normal body temperature. During NMP, the device also allows for ongoing assessment of donor liver function and further viability assessment to help determine suitability of the organ for transplant.
  Interventions: Device: Declined liver in Normothermic Machine Perfusion (NMP)
- Standard cold preservation of liver (Active Comparator): This group will receive liver transplant using the standard method of preservation. There will be 3 comparison groups: one local comparison group and two comparison groups from the national UNOS data.
  Interventions: Procedure: Standard cold preservation of liver

INTERVENTIONS:
Device: Declined liver in Normothermic Machine Perfusion (NMP) — The discarded livers rejected by all other centers and meeting pre-NMP eligibility criteria will receive NMP using the OrganOx® metra device. The NMP-treated liver that meets the viability criteria will be transplanted to patients who are eligible and consented to the study.
  Other Names: NMP-treated livers
  Arms: Declined liver in Normothermic Machine Perfusion (NMP)
Procedure: Standard cold preservation of liver — The study will have three comparison groups - one local comparison group and two comparison groups from the national UNOS data.
  Comparison group 1 will be patients who received a standard liver transplantation and follow-up care at the Washington University/ Barnes Jewish Hospital (n=50). Patients will be matched by a 5-year age category, sex, MELD score, donor liver graft type (e.g., DCD, DBD), donor age (5-year category), and donor sex. Washington University/ Barnes Jewish Hospital maintains a liver transplantation database that prospectively collects pre- and post-transplantation patient data.
  Comparison group 2 will be patients who received DBD liver transplantation in the OPTN/UNOS database (n=100). Patients will be matched by age, sex, MELD score, donor age, and donor sex.
  Comparison group 3 will be patients who received DCD liver transplantation in the OPTN/UNOS database (n=100). Patients will be matched by age, sex, MELD score, donor age, and donor sex.
  Arms: Standard cold preservation of liver

SUMMARY:
This is a prospective, non-randomized, clinical trial of discarded liver transplants that have received normothermic machine perfusion (NMP), compared with standard cold preservation liver transplants. The discarded livers rejected by all other centers and meeting pre-NMP eligibility criteria will receive NMP using the OrganOx® metra device. The NMP-treated liver that meets the viability criteria will be transplanted to patients who are eligible and consented to the study. Liver transplant outcomes will be ascertained during 12 months post-transplantation. The results of the trial will be compared with those of contemporary comparison groups of patients who received the standard criteria donor liver transplantation.

DETAILED DESCRIPTION:
This is a single center, prospective, non-randomized, clinical trial to assess the feasibility of successful transplantation of NMP-treated livers to patients. First, up to 71 marginal livers declined for transplantation will be treated with NMP using the OrganOx® metra device and tested for viability using previously defined criteria. NMP-treated viable livers will be subsequently transplanted to patients (n=5 in the 1st stage; additional 10 transplantation in the 2nd stage; additional 10 transplantation in the 3rd stage: total N=25). Patients will be closely followed for clinical outcomes of the transplantation during 6 months post-transplantation. The follow-up will also be extended up to 1 year post-transplantation. The trial will compare the results to those of three comparison groups - 1) matched patients who received liver transplantation at Washington University/Barnes Jewish Hospital; 2) matched patients who received DBD liver transplantation in the OPTN/UNOS database; and 3) matched patients who received DCD liver transplantation in the OPTN/UNOS database. Given that patient safety is the priority, the trial uses a multi-stage design in which the study stops earlier when NMP-treated liver transplantation is observed to be ineffective (see trial schema in Section 3.1).

ELIGIBILITY:
PRE-NMP DECLINED LIVER ELIGIBILITY:

Inclusion Criteria:

* DCD donor aged 6 years or greater and liver weight between 1 kg and 3.4 kg, with functional warm ischemic time (defined as the period between the systolic blood pressure less than 60 mmHg to the time of commencing donor aortic perfusion) in DCD donors less than 40 minutes
* DCD asystolic warm ischemia time (from heartbeat stopping to initiation of cold flush) less than 15 minutes
* DBD donor aged 6 years or greater and liver weight between 1 kg and 3.4 kg, with less than 8 hours cold ischemia time and DCD livers with less than 7 hours cold ischemia time (defined as the interim from initiation of donor in vivo cold organ preservation to removal of the liver graft from cold storage)
* 'Rapid Recovery' donors for liver procurement, meeting the above criteria
* Suboptimal in situ flush

Exclusion Criteria:

* DBD or DCD donor less than 6 years old
* DCD grafts with donor functional warm ischemic time (defined as the period between the systolic blood pressure less than 60 mmHg to the time of commencing donor aortic perfusion) greater than or equal to 40 minutes
* DCD asystolic warm ischemia time (from heartbeat stopping to initiation of cold flush) greater than or equal to 15 minutes
* DBD livers with cold ischemia time greater than or equal to 8 hours and DCD livers with greater than or equal to 7 hours cold ischemia time
* Donor serum bilirubin greater than or equal to 5 mg/dL
* Liver weight less than 1 kg or greater than or equal to 3.5 kg
* Grafts from patients with HIV infection
* Cirrhotic livers
* Livers with bridging fibrosis

LIVER TRANSPLANTATION - HUMAN

Inclusion criteria:

* Subject must be greater than or equal to 18 years of age.
* Subject with end-stage liver disease who is actively listed for primary liver transplantation on the UNOS waiting list
* Subject, or a legally authorized representative, has given informed consent to participate in the study
* Subject has a frailty classification of "Mild frailty/No frailty (Robust)", based on the Liver Frailty Index (LFI), which has been assessed within 6 months prior to liver transplant OR Subject is able to perform >350 m on a 6 minute walk test (6MWT) within 6 months prior to liver transplant.

  * In all cases, the "most recent" (and within 6 months prior to transplant) measurement of LFI or 6MWT will be used to determine eligibility.

Exclusion criteria:

* Subject is currently listed as a UNOS status 1A.
* Subject is requiring oxygen therapy via ventilator/respiratory support.
* Subject is planned to undergo simultaneous solid organ transplant.
* Subject is pregnant at the time of transplant.
* Subject MELD score 29 or higher
* Subject receives re-transplantation of liver.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2020-12-03 (Actual); Primary Completion 2025-05-14 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of patients with no graft failure at 6 months | Up to 6 months
  6-month graft and patient survival as an indicator of liver function after NMP- treated liver transplantation. 6-month patient survival rate will be estimated as the number of patients who survive by 6 months post-transplantation with NMP-treated livers
  This is a nationally accepted outcome routinely assessed in organ transplantation programs.
  6-month graft survival rate = (Number of patients with no graft failure at 6-month post transplantation)/(Total number patients who received transplantation with NMP-treated liver)
  6-month graft and patient survival rates will be compared to those in each comparison group using Fisher's Exact test.
  Kaplan-Meier survival curve will be examined as well.
Total number of patients who received NMP-treated liver transplantation | Up to 6 months
  6-month patient survival rate will be estimated as the number of patients who survive by 6 months post-transplantation with NMP-treated livers divided by the total number of patients who received NMP-treated liver transplantation.
  6-month patient survival rate = (Number of patients who survive by 6-month post transplantation)/(Total number patients who received transplantation with NMP-treated liver)
  6-month graft and patient survival rates will be compared to those in each comparison group using Fisher's Exact test.
  Kaplan-Meier survival curve will be examined as well.

SECONDARY OUTCOMES:
Assess liver graft function and survival after transplantation | 3 months to 1 year
  Liver graft function assessment: early allograft dysfunction (EAD) and primary non-function (PNF).
  Long-term survivals of patient and graft will provide additional evidence on the safety of using NMP-treated liver for transplantation.
Assess survival after transplantation | 3 months to 1 year
  90-day graft and patient survival
  1-year graft and patient survival
  Long-term survivals of patient and graft will provide additional evidence on the safety of using NMP-treated liver for transplantation.
To assess morbidity associated with receipt of NMP-treated liver | 3 months to 1 year
  1. Incidence of intrahepatic biliary strictures
  2. Incidence of vascular complications
  3. Event rate of requirement of renal replacement therapy
  4. Incidence of biopsy-proven acute rejection
  5. Event rate of transplant related reoperation rate
  6. Length of ICU and hospital stay
  7. Event rate of readmissions and other transplant related serious adverse events
  Incidence rates of adverse outcomes will provide additional evidence on the safety of using previously declined, NMP-treated liver for transplantation
Quality of Life Score Questionnaire | 6 months
  Quality of life score using EQ-5D-5L questionnaire.
  To evaluate the effect of liver transplantation on patient's quality of life. Quality of life questionnaire will be completed at 3 timepoints: Baseline (prior to transplantation), 90 days and month 6
Estimate proportion of declined livers that can be used for transplantation following NMP | 12 months to 18 months
  To estimate the proportion of declined livers that can be used for transplantation following NMP.
  Rescue-rate that is the number of viable NMP- treated livers divided by the total number of NMP-treated livers. The organ recovery rate provides additional evidence on the feasibility of using NMP-treated liver for transplantation.

CONTACTS AND LOCATIONS:
Overall Officials: Will Chapman, MD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Olumba FC, Zhou F, Park Y, Chapman WC; RESTORE Investigators Group. Normothermic Machine Perfusion for Declined Livers: A Strategy to Rescue Marginal Livers for Transplantation. J Am Coll Surg. 2023 Apr 1;236(4):614-625. doi: 10.1097/XCS.0000000000000555. Epub 2023 Jan 11. PMID 36728302